CLINICAL TRIAL: NCT01568294
Title: A Phase 1, Multicenter, Open-label, Dose-escalation Study in Japan to Determine the Tolerated Dose and to Evaluate the Safety, Efficacy, and Pharmacokinetics of Pomalidomide Alone or in Combination With Dexamethasone in Patients With Refractory or Relapsed and Refractory Multiple Myeloma
Brief Title: Japanese Phase 1 Study to Evaluate Tolerated Dose, Safety, and Efficacy of Pomalidomide in Patients With Refractory or Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-004
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pomalidomide (Experimental): Patients will receive pomalidomide orally on Days 1-21 of each 28-day cycle until when/if a discontinuation criterion, e.g., disease progression, development of an unacceptable toxicity, voluntary withdrawal, or pomalidomide is in market for the target indication.
  Interventions: Drug: pomalidomide

INTERVENTIONS:
Drug: pomalidomide — 2 mg or 4mg oral pomalidomide once per day on Days 1-21 of a 28-day cycle

SUMMARY:
The purpose of this study is to determine the tolerated dose of pomalidomide and also to evaluate the pharmacokinetics, safety and efficacy of pomalidomide in patients with refractory or relapsed and refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 20 years of age at the time of signing the informed consent document
* The subject must understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
* Must be able to adhere to the study visit schedule and other protocol requirements
* Subjects must have documented diagnosis of multiple myeloma and have measurable disease
* All subjects must have had at least 2 prior lines of anti-myeloma therapy. Induction therapy followed by stem cell transplant and consolidation/maintenance will be considered as one line
* All subjects must have either refractory or relapsed and refractory disease defined as documented disease progression during or within 60 days of completing their last anti-myeloma therapy.

  * Primary refractory: Subjects who have never achieved any response better than progressive disease (PD) to any previous line of anti-myeloma therapy.
  * Relapsed and refractory: Subjects who have relapsed after having achieved at least stable disease (SD) to at least one prior regimen and then developed progressive disease (PD) on or within 60 days of completing their last anti-myeloma therapy.
* Subjects must have also undergone prior treatment with at least 2 cycles of lenalidomide and at least 2 cycles of bortezomib (either in separate regimens or within the same regimen).
* All subjects must have received adequate prior alkylator therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.

Exclusion Criteria:

* Pregnant or breastfeeding females
* Hypersensitivity to thalidomide, lenalidomide, or dexamethasone
* ≥ Grade 3 rash during prior thalidomide or lenalidomide therapy
* Patients unable or unwilling to undergo antithrombotic prophylactic treatment will not be eligible to participate in this study
* Any of the following laboratory abnormalities:

  * Absolute neutrophil count (ANC) < 1,000/µL
  * Platelet count < 75,000/µL for patients in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count < 30,000/µL for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells
  * Creatinine Clearance < 45 mL/min according to Cockcroft-Gault formula
  * Corrected serum calcium > 14 mg/dL (> 3.5 mmol/L)
  * Hemoglobin < 8 g/dL (< 4.9 mmol/L; prior RBC transfusion or recombinant human erythropoietin use is permitted)
  * Serum glutamic oxaloacetic transaminase (SGOT) /aspartate aminotransferase (AST) or serum glutamic pyruvic transaminase (SGPT) /alanine aminotransferase (ALT) > 3.0 x upper limit of normal (ULN)
  * Serum total bilirubin > 2.0 mg/dL (34.2 μmol/L); or ≥ 3.0 x upper limit of normal (ULN) for subjects with hereditary benign hyperbilirubinaemia
* Peripheral neuropathy ≥ Grade 2
* Patients who received any of the following within the last 14 days of initiation of study treatment:

  * Plasmapheresis
  * Major surgery (kyphoplasty is not considered major surgery)
  * Radiation therapy
  * Use of any anti-myeloma drug therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2015-07-08 (Actual); Study Completion 2015-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity in accordance with Common Terminology Criteria for Adverse Events | Up to 28 Days
  Incidence of dose-limiting toxicity in accordance with Common Terminology Criteria for Adverse Events

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 28 days
  Maximum observed plasma concentration (Cmax)
Time to maximum observed plasma concentration (tmax) | Up 28 days
  Time to maximum observed plasma concentration (tmax)
Area under the plasma concentration-time curve (AUC0-t) | Up to 28 days
  Area under the plasma concentration-time curve (AUC0-t)
Apparent total plasma clearance (CL/F) | Up to 28 days
  Apparent total plasma clearance (CL/F)
Apparent total volume of distribution (Vz/F) | Up to 28 days
  Apparent total volume of distribution (Vz/F)
Estimate of the terminal elimination half-life in plasma (t1/2) | Up to 28 days
  Estimate of the terminal elimination half-life in plasma (t1/2)
Safety (the number of participants with adverse events, incidence, severity, causality) | Up to 2 years
  Safety (the number of participants with adverse events, incidence, severity, causality)
Progression-free survival | Up to 28 days
  Progression-free survival
Myeloma response | Up to 28 days
  Myeloma response
Time to Response | Up to 28 days
  Time to Response
Duration of Response | Up to 28 days
  Duration of Response

CONTACTS AND LOCATIONS:
Overall Officials: Toru Sasaki, Study Director — Celgene K.K
Locations (8):
- Japan (8):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Tokai University Hospital, Isehara, Kanagawa
  - Saitama Medical Center, Saitama Medical University, Kawagoe, Saitama
  - National Cancer Center Hospital, Tyuuou, Tokyo
  - Kyusyu University Hospital, Fukuoka
  - Kameda General Hospital, Kamogawa
  - Niigata Cancer Center Hospital, Niigata
  - Okayama Medical Center, Okayama

REFERENCES:
- [Background] Matsue K, Iwasaki H, Chou T, Tobinai K, Sunami K, Ogawa Y, Kurihara M, Midorikawa S, Zaki M, Doerr T, Iida S. Pomalidomide alone or in combination with dexamethasone in Japanese patients with refractory or relapsed and refractory multiple myeloma. Cancer Sci. 2015 Nov;106(11):1561-7. doi: 10.1111/cas.12772. Epub 2015 Nov 4. PMID 26292221
- [Background] Mark TM, Forsberg PA, Rossi AC, Pearse RN, Pekle KA, Perry A, Boyer A, Tegnestam L, Jayabalan D, Coleman M, Niesvizky R. Phase 2 study of clarithromycin, pomalidomide, and dexamethasone in relapsed or refractory multiple myeloma. Blood Adv. 2019 Feb 26;3(4):603-611. doi: 10.1182/bloodadvances.2018028027. PMID 30792190